CLINICAL TRIAL: NCT01154673
Title: Randomized, Double-blinded, Controlled Trial of Intensive HAART Including Raltegravir, and Maraviroc, on HIV-1 Pro-viral DNA and Reservoir Decay in HIV-1-infected Individuals During the Acute/Early Infection
Brief Title: Effects of Intensive cART During Acute/Early HIV Infection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Unity Health Toronto (Other); Maple Leaf Research (Other)
Responsible Party: Principal Investigator, Mario Ostrowski, Principal Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 041009; NCT01101516 (obsolete NCT alias)
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Acute HIV Infection
MeSH Terms: interventions — Raltegravir Potassium; Maraviroc; Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Lopinavir; Ritonavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive HAART (Experimental): Patients in this arm will receive the following HAART regimen:
  Raltegravir 400 mg BID + Maraviroc 150mg BID + emtricitabine 200mg /tenofovir 300mg QD + lopinavir 400 mg/ritonavir 100mg BID for 96 weeks
  Interventions: Drug: raltegravir; Drug: maraviroc; Drug: emtricitabine 200mg /tenofovir 300mg; Drug: lopinavir 400 mg/ritonavir 100mg
- Placebo Arm (Placebo Comparator): Placebo (in place of raltegravir and maraviroc) will be added to standard HAART (Emtricitabine 200mg /tenofovir 300mg QD + Lopinavir 400 mg/ritonavir 100mg BID) for 48 weeks and then offered open label Raltegravir and Maraviroc after 48 weeks
  Interventions: Drug: emtricitabine 200mg /tenofovir 300mg; Drug: lopinavir 400 mg/ritonavir 100mg

INTERVENTIONS:
Drug: raltegravir — Raltegravir 400 mg BID + Maraviroc 150mg BID in addition to standard HAART
  Other Names: Isentress; MK-0518
  Arms: Intensive HAART
Drug: maraviroc — Raltegravir 400 mg BID + Maraviroc 150mg BID in addition to standard HAART
  Other Names: Celsentri; Selzentry
  Arms: Intensive HAART
Drug: emtricitabine 200mg /tenofovir 300mg — emtricitabine 200mg /tenofovir 300mg QD
  Other Names: Truvada
Drug: lopinavir 400 mg/ritonavir 100mg — lopinavir 400 mg/ritonavir 100mg BID
  Other Names: Kaletra; Aluvia

SUMMARY:
This trial will investigate the efficacy and safety of intensified antiretroviral treatment that includes raltegravir and maraviroc during the early stages of HIV infection. With the proven efficacy of these antiviral drugs in pre- and post-clinical trials, we would like to investigate the ability of the combination of raltegravir and maraviroc plus a standard HAART backbone to further decrease the viral load in acutely infected treated HIV infected individuals.

DETAILED DESCRIPTION:
The trial is a prospective, randomized, double-blinded, placebo-controlled study with follow-up to 5 years. Thirty-two individuals presenting with newly diagnosed acute or early HIV-1 infection as described in the inclusion criteria will be enrolled, with sixteen randomized to each arm. Individuals will be randomized to one of two arms: the "Intensive" arm with standard HAART (Emtricitabine 200mg /tenofovir 300mg QD + Lopinavir 400mg /ritonavir 100mg BID) + Raltegravir + Maraviroc or the "placebo" arm with standard HAART+ Placebo for 48 weeks. Another group of individuals diagnosed with acute or early HIV-1 who elect to forego early treatment will be followed as non-randomized, untreated controls. At week 48, all patients will be informed of study results. If results are positive in the intensive treatment group, the placebo group will be offered to roll-over to the intense treatment arm and followed as an open-label cohort out to five years. Participants may stop treatment at any time and withdraw from the study. If they choose to do so, they will be followed according to the standards employed for all HIV-1 patients at the Maple Leaf clinic. At the five year point, the decision to terminate treatment will be made based on the existing state of the HIV-1 literature at the time.

ELIGIBILITY:
Inclusion Criteria:

The major single criterion for inclusion into the study will be the presence of confirmed acute/early HIV-1 infection, as defined by one of the three following criteria:

1. Positive HIV-1 antibody test result (Western blot), with a documented negative test result in the previous six months or
2. Positive or weakly positive HIV-1 antibody screening ELISA test result, with indeterminate and evolving confirmatory test result with demonstrated HIV-1 antigenemia (p24 antigen test result) or viremia (HIV-1 bDNA ≥ 500 copies/ml) or
3. Negative HIV-1 antibody test result in the setting of an illness compatible with acute seroconversion with demonstrated HIV-1 antigenemia (p24 antigen test result) or plasma viremia (HIV-1 bDNA ≥ 500 copies/ml)

Other inclusion criteria are:

* Ages 18 or older
* Ability to provide informed consent
* HIV-1 viral load ≥ 5,000 copies/ml

Exclusion Criteria:

1. Participants who would have difficulty participating in a trial due to non-adherence or substance abuse
2. Participants with any of the following abnormal laboratory test results in screening:

   * Hemoglobin < 85 g/L
   * Neutrophil count < 750 cells/uL
   * Platelet count < 50,000 cells/L
   * AST or ALT > 5X the upper limit of normal
   * Creatinine > 250 umol/L
3. Participant with a malignancy
4. Participant with other significant underlying disease (non-HIV-1) that might impinge upon disease progression or death
5. Participant who is pregnant or who is trying to conceive

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Ostrowski, MD, Principal Investigator — University of Toronto; Colin Kovacs, MD, Principal Investigator — Maple Leaf Research
Locations (2):
- Canada (2):
  - University of Toronto, Toronto, Ontario
  - Maple Leaf Medical Clinic, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensive HAART: Patients in this arm will receive the following HAART regimen:
  Raltegravir 400 mg BID + Maraviroc 150mg BID + emtricitabine 200mg /tenofovir 300mg QD + lopinavir 400 mg/ritonavir 100mg BID and endpoint is measured at 48 weeks
- Placebo Arm: Placebo (in place of raltegravir and maraviroc) will be added to standard HAART (Emtricitabine 200mg /tenofovir 300mg QD + Lopinavir 400 mg/ritonavir 100mg BID) and endpoint is measured at 48 weeks
Period: Overall Study
Arm/Group | Intensive HAART | Placebo Arm
Started | 16 | 16
Completed | 14 | 16
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — moved out of province | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intensive HAART: Patients in this arm will receive the following HAART regimen:
  Raltegravir 400 mg BID + Maraviroc 150mg BID + emtricitabine 200mg /tenofovir 300mg QD + lopinavir 400 mg/ritonavir 100mg BID
- Placebo Arm: Placebo (in place of raltegravir and maraviroc) will be added to standard HAART (Emtricitabine 200mg /tenofovir 300mg QD + Lopinavir 400 mg/ritonavir 100mg BID)
- Total: Total of all reporting groups
Arm/Group | Intensive HAART | Placebo Arm | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 34 [22 to 59] | 30 [23 to 49] | 32 [22 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 16 | 32
Region of Enrollment [Number; unit: participants]
  Canada | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in Proviral HIV-1 DNA in Total CD4+ T-cells From Baseline to Week 48 in Participants Randomized to the Intensified Arm Versus the Control Arm Who Received Placebo in Addition to Standard HAART.
Description: The level of HIV Provirus in CD4 T cells obtained from peripheral blood at 48 weeks compared to baseline. A quantitative HIV PCR assay was done. The mean/median values from the standard HAART group is compared to the intensive HAART treatment regimen.
Time Frame: Baseline to Week 48
Measure: Median (Full Range); unit: HIV DNA copies/ million CD4 cells
Arm/Group | Intensive HAART | Placebo Arm
Number analyzed (Participants) | 14 | 16
HIV DNA copies/ million CD4 cells | 279 [26 to 2836] | 244 [2.5 to 5186]
Statistical Analysis 1: Comparison: Intensive HAART vs Placebo Arm; Test type: Superiority or Other; p = 0.056, Regression, Linear — "The estimated difference in mean change from baseline to 48 weeks was calculated as the log DNA copies/106 CD4+ T cells in "Intensive HAART" minus the log DNA copies/106 CD4+ T cells in "Placebo Arm"; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-.006 to 0.4] — The estimated difference in mean change from baseline to 48 weeks was calculated as the log DNA copies/106 CD4+ T cells in "Intensive HAART" minus the log DNA copies/106 CD4+ T cells in "Placebo Arm"

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Intensive HAART | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive HAART (N=16) | Placebo Arm (N=16)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — one participant experience unexpected neutropenia after the primary endpoint of 48 weeks, which was transient and resolved and was felt to be due to other medications the participant was taking rather than the study medications by the investigators.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No